CLINICAL TRIAL: NCT07207954
Title: A Phase 1a/1b, Randomized, Double-Blind, Placebo- and Active-Controlled, Single and Multiple Ascending Dose Study Evaluating the Comparative Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LFD-200 in Adult Participants Who Are Healthy or Have Moderate to Severe Rheumatoid Arthritis
Brief Title: Study of LFD-200 in Healthy Adults and Adults With Moderate to Severe Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lifordi Immunotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LFD200A11
Record Dates: First submitted 2025-09-19; First posted 2025-10-06 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; Rheumatoid Arthritis; Healthy Participants; Phase 1a/1b; Safety; Tolerability; Pharmacokinetics; Pharmacodynamics; First in human; Single Ascending Dose; Multiple Ascending Dose
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: SAD in HP (Experimental): Three planned cohorts (SAD HP Cohorts 1 to 3) and 3 optional cohorts (SAD HP Cohorts 4 to-6) of 11 participants each will receive a single SC dose of LFD-200, a single SC dose of matching saline placebo, or a single oral dose of open label 10 mg prednisone. Within each cohort, 6 participants will be randomly assigned to receive LFD-200, 2 participants will receive saline placebo, and 3 will receive prednisone.
  Interventions: Drug: LFD-200; Other: Placebo; Drug: Oral Prednisone
- Part 1: MAD in HP (Experimental): Two planned cohorts (MAD HP Cohorts 1 and 2) of 8 HPs each (16 total) will be randomly assigned to receive 4 weekly SC doses of LFD-200 (6 participants) or saline placebo (2 participants) over a duration of 22 days.
  Interventions: Drug: LFD-200; Other: Placebo
- Part 2: MAD in RA (Experimental): Two planned cohorts (MAD RA Cohorts 1 and 2) of 14 RA participants each (28 total) will be randomly assigned to receive either up to 13 weekly SC doses of LFD-200 over 85 days with a daily prednisone placebo tablet (LFD-200 arm; 8 participants), or up to 13 weekly SC doses of saline placebo over 85 days with daily prednisone placebo tablet (placebo arm; 3 participants), or up to 13 weekly SC doses of saline placebo over 85 days with a daily dose of oral prednisone (prednisone arm; 3 participants)
  Interventions: Drug: LFD-200; Other: Placebo; Drug: Oral Prednisone

INTERVENTIONS:
Drug: LFD-200 — 2 mL glass vials, as 150 mg/mL concentrated solution
Other: Placebo — 0.9% NaCl
Drug: Oral Prednisone — Tablet
  Arms: Part 1: SAD in HP; Part 2: MAD in RA
Other: Placebo — Placebo tablet to match Prednisone
  Arms: Part 2: MAD in RA

SUMMARY:
This is a double-blind, randomized, placebo- and active-controlled study investigating the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of subcutaneous (SC) doses of LFD-200. The study design includes: a single ascending dose (SAD) study in up to 66 adult healthy participants (HPs) to investigate the effects of a single SC dose, with a 30-day follow-up; a multiple ascending dose (MAD) study in up to 40 HPs to assess up to 4 weekly SC doses, with a 30-day follow-up after the last dose; and a MAD study in up to 70 participants with moderate to severe rheumatoid arthritis (RA) to evaluate up to 13 weekly SC doses, with a 30-day follow-up after the last dose.

ELIGIBILITY:
Inclusion Criteria for Healthy Participants:

* Age 18-55
* BMI - 18-32
* Participants must be deemed by the Investigator to be generally healthy individuals based on a medical evaluation that includes a physical examination, medical history, vital signs, and the results from clinical labs and other safety assessments collected during the Screening period.

Exclusion Criteria for Healthy Participants:

* Participants with any current or previous illness that, in the opinion of the investigator, might confound the results of the study or pose an additional, unacceptable risk to the participant or that could prevent, limit, or confound the protocol specified assessments or study results' interpretation.
* Recent serious or ongoing infection
* Known/suspected primary immunodeficiency
* Receipt of injected or systemic glucocorticoids within 6 weeks prior to screening
* Use of prohibited medications
* Any of the following lab abnormalities:

  * White blood cell (WBC) count <3.0 x 109/L
  * Absolute neutrophil count (ANC) <2.0 x 109/L
  * Hemoglobin (Hgb) <12.5 g/dL for males and <11.5 g/dL for females
  * Platelet count <140 x 109/L
  * Alanine transaminase (ALT) ≥1.2x upper limit of normal (ULN)
  * Total bilirubin ≥1.2x ULN (except if Gilbert's disease is suspected etiology)
  * Estimated glomerular filtration rate (eGFR) <80 mL/min/1.73m2 based on Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI 2021) formula.
  * International normalized ratio (INR) ≥1.2 × ULN
  * Glycated hemoglobin (HbA1c) >6%
  * Positive urine cotinine test (Day -1 only), alcohol breath test or urine drug screen for substances of abuse. Positive tetrahydrocannabinol (THC) is not exclusionary.
  * A Screening thyroid stimulating hormone (TSH) level that is <0.9 × lower limit normal (LLN) or ≥1.2 × ULN
  * Cortisol level <1.0 × LLN (Collected in the AM at the Baseline Visit)

Inclusion Criteria for RA Participants:

* Adults of age 18 to 75 years, inclusive, at the time of signing the ICF.
* BMI within the range of 18.0- to 35.0 kg/m² (inclusive).
* Has RA for ≥6 months.
* Positive rheumatoid factor (RF) or anti-citrullinated protein antibody (ACPA) test at Screening (low or high positive acceptable).
* A high-sensitivity C-reactive protein (hsCRP) level at Screening must be >ULN.
* Has active RA disease defined as follows:

  * Disease Activity Score of 28 joints-CRP (DAS28-CRP) >3.2 at Screening and Baseline
  * Has ≥4 swollen and ≥4 tender joints on a 28-joint count at Screening and Baseline
* On MTX orally or subcutaneously for at least 12 weeks prior to Screening. Dose of MTX (including route of administration) must have been stable at 15 to 25 mg weekly (or 10 to15mg in case of documented intolerance) for ≥ 12weeks at Randomization with plans to continue it at the same dose and route of administration for the duration of the study.

Exclusion Criteria for RA Participants:

* Clinical evidence of significant unstable or uncontrolled acute or chronic diseases (e.g., cardiac [including congestive heart failure, angina, or history of myocardial infarction], pulmonary [including chronic obstructive pulmonary disease, asthma requiring systemic GC therapy, pulmonary hypertension, or pulmonary fibrosis], hematologic, gastrointestinal, hepatic, renal, neurological, psychiatric, dermatologic, musculoskeletal, or infectious diseases) that, in the opinion of the Investigator or Sponsor, constitutes an inappropriate risk or contraindication for participation in study or that could interfere with study objectives, conduct, or evaluation
* Any other autoimmune or autoinflammatory disorder, which in the opinion of Investigator/Sponsor would constitute an inappropriate risk or a contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation.
* Recent serious or ongoing infection, or risk for serious infection, or acute or chronic infection
* Known seropositivity for or active infection by HIV or strongyloides (if at risk of exposure (e.g., travel from/reside in endemic area))
* Active or latent TB infection, as suggested by a positive chest radiograph OR positive/indeterminate QFT-TB Gold Plus or T-SPOT within the 12 weeks prior to Screening or a positive Screening CXR or QFT test. Indeterminate screening QFT tests are also exclusionary but may be repeated once and will be considered positive if retest results are positive or indeterminate/borderline.
* Clinically significant abnormalities on ECG per the Investigator or Sponsor or any of the following mean ECG parameters on screening/baseline (triplicate) ECG:

  * HR <40 or >100 beats per minute
  * QTcF (Fridericia corrected QT) interval >450 ms (males) or >470 ms (females)
  * QRS interval >120 ms
  * PR interval >220 ms
* Use or anticipated use of medications for the timeframes specified below:

  * Unstable use of any herbal medicines (e.g., St. John's wort) and supplements within 4 weeks prior to Screening through Baseline or anticipated changes in use during study.
  * Systemic or local (e.g., topical, oral, ophthalmic) corticosteroid (CS) use within 6 weeks prior to randomization or anticipated use during the study (other than as study intervention).
  * Any intra-articular injection within 4 weeks prior to Screening through Baseline or anticipated use during the study.
  * Use of cyclophosphamide, chlorambucil, leflunomide for <6 months or cyclosporine, mycophenolic acid, azathioprine, tacrolimus, or gold <8 weeks prior to Screening through Baseline or anticipated use during the study.
  * Receipt of rituximab or any other cell depleting biologic therapy within 1 year of Screening through Baseline or anticipated use during the study.
  * Use of any other commercial injectable biologic (including those for other non- arthritic conditions such as asthma, osteoporosis, lipids, atopic dermatitis) within 12 weeks or 5 half-lives (whichever is longer) prior to Screening through Baseline, or anticipated use during the study.
  * Use of any other oral DMARD, including JAK-inhibitors, within 12 weeks prior to Screening through Baseline or anticipated used during the study. MTX or HCQ use is permitted as specified in the Inclusion Criteria
  * Use of >1 systemic biologic therapy for the treatment of RA prior to Screening or Baseline. For those participants that have used no more than one systemic biologic therapy, the systemic biologic therapy must have been discontinued at least 12 weeks or 5 half-lives (whichever is longer) prior to Screening with no use through Baseline or anticipated use during the study.
  * Receiving or has received any investigational drug (or is currently using an investigational device) within 30 days or 5 half-lives (whichever is longer), prior to Screening.
  * Unstable use of topical or systemic nonsteroidal anti-inflammatory drugs (NSAIDs) OR use above the maximum allowed doses OR use of more than 1 systemic NSAID (other than prophylactic aspirin ≤325mg daily) in the 2 weeks prior to Screening through Baseline or anticipated use during the study.
* The presence at Screening of any laboratory values of concern in the opinion of the Investigator or Sponsor or of any of the below based on central laboratory testing at Screening:

  * WBC count <3.0 × 10⁹/L
  * ANC <2.0 × 10⁹/L
  * Hgb <10 g/dL
  * Platelet count <100 × 10⁹/L
  * ALT >2 × ULN
  * Total bilirubin ≥1.5 × ULN (unless Gilbert's disease is suspected)
  * eGFR <45 mL/min/1.73m² estimated based on CKD-EPI 2021 formula
  * International normalized ratio >1.2 × ULN
  * HbA1c >8%
  * AM cortisol level at Baseline Visit <0.9 × LLN
  * Positive alcohol breath test or urine drug screen for substances of abuse. Positive THC or positivity for other substances due to ongoing use of these drugs under physician supervision (e.g., prescription narcotics for known pain disorder) are not exclusionary.
  * A Screening TSH level that is <0.9 × LLN or > 1.1 × ULN.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-07-16 (Estimated); Study Completion 2027-07-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Baseline up to 30 days after last dose.
  Number of participants experiencing any adverse events during the study period.
Severity of Adverse Events (AEs) | Baseline up to 30 days after last dose.
  Classification of adverse events based on severity (mild, moderate, severe).
Seriousness of Adverse Events (AEs) | Baseline up to 30 days after last dose.
  Number of participants experiencing serious adverse events (SAEs) during the study period.
Change from Baseline in Blood Pressure (BP) | Baseline up to 30 days after last dose.
  Difference in systolic and diastolic blood pressure measurements from baseline to specified time points.
Change from Baseline in Temperature | Baseline up to 30 days after last dose.
  Difference in body temperature measurements from baseline to specified time points.
Change from Baseline in Respiratory Rate | Baseline up to 30 days after last dose.
  Difference in respiratory rate measurements from baseline to specified time points.
Change from Baseline in Heart Rate (HR) | Baseline up to 30 days after last dose.
  Difference in heart rate measurements from baseline to specified time points.
Change in Hemeglobin from Baseline to specified timepoints | Baseline up to 30 days after last dose.
  Hemeglobin is measured in g/dL
Change in Alanine Aminotransferase from Baseline to specified timepoints | Baseline up to 30 days after last dose.
  Alanine Aminotransferase is measured in U/L
Change in Leukocytes in urine from Baseline to specified timepoints | Baseline up to 30 days after last dose.
  Leukocytes in urine is measured in x10^6/L
Change in Heart Rate (HR) from Baseline to specified timepoints | Baseline up to 30 days after last dose.
  Heart rate is measured in beats per minute
Change from Baseline in PR Interval | Baseline up to 30 days after last dose.
  Difference in PR interval measurements from baseline to specified time points.
Change from Baseline in QRS Interval | Baseline up to 30 days after last dose.
  Difference in QRS interval measurements from baseline to specified time points.
Change from Baseline in QT Interval | Baseline up to 30 days after last dose.
  Difference in QT interval measurements from baseline to specified time points.
Primary Outcome Measure: Change from Baseline in QTcF Interval | Baseline up to 30 days after last dose.
  Difference in QTcF interval measurements from baseline to specified time points.
Incidence of Clinical Findings on Physical Examination | Baseline up to 30 days after last dose.
  Number of participants with clinical findings during physical examinations, including injection site reactions.
Severity of Clinical Findings on Physical Examination | Baseline up to 30 days after last dose.
  Classification of clinical findings based on severity (mild, moderate, severe), including injection site reactions.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Baseline up to 30 days after last dose.
  The highest concentration of the drug observed in plasma after administration.
Trough Concentration (Ctrough) | Baseline up to 30 days after last dose.
  The lowest concentration of the drug observed in plasma before the next dose.
Average Concentration (Cavg) | Baseline up to 30 days after last dose.
  The average concentration of the drug in plasma over a specified time period
Clearance | Baseline up to 30 days after last dose.
  The rate at which the drug is removed from the body.
Volume of Distribution | Baseline up to 30 days after last dose.
  The volume in which the drug is distributed in the body.
Area Under the Plasma Concentration vs. Time Curve from Time Zero to the Last Quantifiable Concentration (AUClast) | Baseline up to 30 days after last dose.
  The area under the plasma concentration-time curve from the time of dosing to the last measurable concentration.
Area Under the Plasma Concentration vs. Time Curve from Time Zero Extrapolated to Infinity (AUCinf) | Baseline up to 30 days after last dose.
  The area under the plasma concentration-time curve from the time of dosing extrapolated to infinity.
Area Under the Plasma Concentration vs. Time Curve from Time Zero to 168 Hours Post-Dose (AUC0-168) | Baseline up to 30 days after last dose.
  The area under the plasma concentration-time curve from the time of dosing to 168 hours post-dose.
Area Under the Plasma Concentration vs Time Curve Over the Dosing Interval (AUCtau) | Baseline up to 30 days after last dose.
  The area under the plasma concentration-time curve over the dosing interval.
Accumulation Ratio (Rac) | Baseline up to 30 days after last dose.
  The ratio of drug accumulation in plasma after multiple dosing compared to a single dose.
Time Corresponding to the Maximum Observed Plasma Concentration (Tmax) | Baseline up to 30 days after last dose.
  The time at which the maximum plasma concentration of the drug is observed.
Change from Baseline in Cortisol Levels | Baseline up to 30 days after last dose.
  Difference in cortisol levels from baseline to specified time points.
Change from Baseline in Bone Biomarkers | Baseline up to 30 days after last dose.
  Difference in Bone Biomarker levels from baseline to specified time points
Change from Baseline in DAS28-CRP | Baseline up to 30 days after last dose.
  Difference in Disease Activity Score 28 - C-reactive protein (DAS28-CRP) from baseline to specified time points for rheumatoid arthritis (RA) cohorts.

CONTACTS AND LOCATIONS:
Locations (6):
- Nucleus Network, Melbourne, Australia
- Clinical Republican Hospital "Timofei Mosneaga", ARENSIA E.M., Chisinau, Moldova
- Poland (3):
  - MICS Centrum Medyczne Torun - MICS - PPDS, Torun
  - National Institute of Geriatrics, Rheumatology and Rehabilitation, Warsaw, Poland, Warsaw
  - Centrum Medyczne Reuma Park, Warsaw
- "ARENSIA EXPLORATORY MEDICINE" LIMITED LIABILITY COMPANY, Medical Center, Department of Clinical Trials, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No